CLINICAL TRIAL: NCT06538363
Title: Running Online Injury Prevention Feasibility Study
Acronym: ROIPF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Principal Investigator, Chris Napier, Assistant Professor, Simon Fraser University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SimonFraserU
Record Dates: First submitted 2024-07-25; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Musculoskeletal Injury
Keywords: Running; Wearable sensors; Biomechanics; Training; Education; Female athlete
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Control and Intervention group
Who Masked: Participant
Masking Description: Participants will be blinded to their group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Behavioral: Generic Education
- Intervention (Experimental)
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Personalized training advice
  Arms: Intervention
Behavioral: Generic Education — Generic training advice
  Arms: Control

SUMMARY:
The main purpose of this study is to test the feasibility of a larger scale interventional study. The investigators want to understand whether data can be reliably collected data various different streams while participants follow a standard 12-week half-marathon training program, and whether participants follow training recommendations.

DETAILED DESCRIPTION:
Research procedures will include an online eligibility questionnaire, a demographic intake questionnaire, a weekly injury questionnaire, and an exit questionnaire (hosted on the SFU Survey Monkey platform). This study involves an initial in-person 1-hour orientation session. Multiple dates will be offered in order to accommodate participants. Participants will be randomly allocated to either the control or intervention group. All participants will be given a pair of running shoes (Hettas Sport Ltd.). Half of the participants in each group will also be outfitted with a pair of shoe-embedded sensors (Plantiga Technologies, Inc.). All participants will also be given access to a menstrual cycle tracking app (MyNormative). If participants have a Strava profile already, this will be linked to the study third-party data extraction API called "Strava API" to give the research team access to select workout data. If participants do not have a Strava profile, an anonymous profile will be created and linked to the API. Participants will be oriented on how to use the shoe-embedded sensors and MyNormative app. Following a one to two week familiarization period in which the participants can become comfortable with the protocol, participants will commence a 12-week half-marathon training program guided by a coach. The training program will consist of four runs per week, including two optional in-person group runs, and will culminate with a half-marathon race. Over the course of the training program, participants will be responsible for uploading the data from the shoe-embedded sensors after each run (for those that have them), tracking their menstrual cycle with the MyNormative app, and recording their runs with their GPS-enabled smartwatch which will automatically upload training data to Strava. Participants in the intervention group will be given individualized training recommendations based on their training data uploaded to Strava (e.g., "Training load is high, take a rest day tomorrow" or "Training load is appropriate, continue as planned"). Training load will be calculated from average distance, speed, step count, and heart rate. Participants in the control group will receive generic training recommendations (e.g., "Keep up the good work" or "Make sure to balance training with enough recovery time"). Communication with the participants will occur via text message on their personal cell phone. Following completion of the study, participants in the intervention group will be asked to complete an online questionnaire about why the participants did/did not follow the individualized training advice. Participants will be permitted to keep the running shoes but will be required to return the shoe-embedded sensors at study completion.

ELIGIBILITY:
Inclusion Criteria:

* Cis-gender female (someone who was born female and currently identifies as a woman) runners
* Over the age of 18
* Have not been injured in the last 3 months (**For the purpose of this study, an injury is defined as "musculoskeletal (originating from the bones, muscles, joints) that has restricted the ability to run in any way (distance, speed, duration) for at least 7 days or for 3 consecutive training sessions"**)
* Have run on average 3 times/week for the last 6 months
* Own a GPS-enabled smart watch with an optical wrist heart rate sensor
* Fit shoe size between 6.5 and 8.5 US women's sizing
* Able to attend one of the in-person orientation sessions
* Able to understand written and spoken English

Exclusion Criteria:

* Any current pain with running

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gender females
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | 4 weeks
  - The number of participants enrolled versus the target number.
Data Collection Compliance | 12 weeks
  * The percentage of participants who complete the online eligibility questionnaire, demographic intake questionnaire, weekly injury questionnaire, and exit questionnaire.
  * The percentage of participants who reliably upload data from the shoe-embedded sensors after each run.
  * The percentage of participants who consistently track their menstrual cycle with the MyNormative app.
  * The percentage of participants who regularly record their runs with their GPS-enabled smartwatch and upload data to Strava.
Attendance | 16 weeks
  - Attendance rate at the initial in-person orientation session and optional in-person group runs.
Adherence to Training Recommendations | 12 weeks
  - Percentage of participants in the intervention group who follow the individualized training recommendations.
Training Program Compliance | 12 weeks
  - Percentage of completed prescribed training runs per week during the 12-week half-marathon training program.
Satisfaction and Usability | 12 weeks
  * Participant feedback on the ease of use and satisfaction with the shoe-embedded sensors, MyNormative app, and Strava integration. Measured during the exit questionnaire.
  * Participant feedback on the clarity and usefulness of the training recommendations (both individualized and generic). Measured during the exit questionnaire.
Barriers and Facilitators | 12 weeks
  - Reasons provided by participants in the intervention group for following or not following the individualized training advice, as captured in the exit questionnaire.

SECONDARY OUTCOMES:
Injury incidence | 12 weeks
  - Incidence and severity of running-related injuries reported weekly via the injury questionnaire. Injuries are defined according to the consensus definition of running injuries by Yamato et al ("musculoskeletal (originating from the bones, muscles, joints) that has restricted your ability to run in any way (distance, speed, duration) for at least 7 days or for 3 consecutive training sessions").

CONTACTS AND LOCATIONS:
Overall Officials: Chris Napier, PhD, Principal Investigator — Simon Fraser University
Locations (1):
- Simon Fraser University, Burnaby, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yamato TP, Saragiotto BT, Lopes AD. A consensus definition of running-related injury in recreational runners: a modified Delphi approach. J Orthop Sports Phys Ther. 2015 May;45(5):375-80. doi: 10.2519/jospt.2015.5741. Epub 2015 Mar 26. PMID 25808527